CLINICAL TRIAL: NCT04982302
Title: Evaluation of Salivary and Intestinal Microbiological Response in Patients With Stage III-IV Periodontitis After Non-surgical Periodontal Therapy
Brief Title: Gut Microbial Changes After Periodontal Treatment
Status: Completed | Type: Observational
Sponsor: University of Turin, Italy (Other)
Responsible Party: Sponsor
Other Study IDs: Perio-gut connection
Record Dates: First submitted 2021-07-19; First posted 2021-07-29 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2022-10

CONDITIONS: Periodontitis; Dysbiosis; Intestinal Disease
MeSH Terms: conditions — Periodontitis; Dysbiosis; Intestinal Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Saliva and stool samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Non-surgical periodontal treatment NSPT: Subgingival instrumentation with ultrasonic devices and curettes of all periodontal pockets in 2 or 4 appointments
  Interventions: Procedure: Non-surgical periodontal treatment

INTERVENTIONS:
Procedure: Non-surgical periodontal treatment — Subgingival instrumentation with ultrasonic devices and curettes of all periodontal pockets

SUMMARY:
Periodontitis is a chronic inflammatory disease of the tooth supporting structures induced by a dysbiosis in the oral and subgingival microenvironment of susceptible patients. The long-term swallowing of high doses of periodontal pathogenic microorganisms could induce a dysbiosis of the intestinal microbiota, favouring the establishment of an 'inflamed' microbiome in terms of composition and/or function. The present project is aimed at a better understanding of the etiopathogenetic correlation between periodontitis and intestinal dysbiosis, and aims to explore the hypothesis that non-surgical periodontal treatment may reduce bacterial alpha diversity in stool samples. Fifty patients affected by stage III-IV periodontitis will be recruited, and treated by means of full-mouth scaling and root planing. Salivary and stool samples, together with a complete periodontal charting and a food diary will be collected and compared at baseline and 3 months after treatment. Age, gender and BMI-matched healthy individuals will be recruited as controls.

ELIGIBILITY:
Inclusion Criteria:

* periodontitis Stage III or IV
* BMI between 20 and 29 kg/m2
* free diet
* presence of at least 20 teeth

Exclusion Criteria:

* systemic diseases (including diabetes, thyroid, liver, or kidney diseases)
* dietary allergies
* use of antibiotics or probiotics during the previous 30 days
* pregnancy or breast feeding

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Study population will be consecutively selected among the patients diagnosed of Stage III-IV periodontitis at the Section of Periodontology of the C.I.R. Dental School of Turin.
Sampling Method: Non-Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Changes in microbiome alpha diversity measured from stool samples at 3 months | [Time Frame: Baseline and 90 days]
  Taxonomic and functional variation of gut bacteria after treatment

SECONDARY OUTCOMES:
Changes in microbiome alpha diversity measured from saliva samples at 3 months | [Time Frame: Baseline and 90 days]
  Taxonomic and functional variation of salivary bacteria after treatment
Changes in mean clinical attachment level (CAL) at 3 months | [Time Frame: Baseline and 90 days]
  Variation in CAL after therapy assessed using a millimetre marked manual periodontal probe at 6 sites per tooth element
Changes in periodontal pocket depth (PPD) at 3 months | [Time Frame: Baseline and 90 days]
  Variation in PPD after therapy assessed using a millimetre marked manual periodontal probe at 6 sites per tooth element
Changes in full mouth bleeding score (FMBS) at 3 months | [Time Frame: Baseline and 90 days]
  Variation in the percentage of bleeding sites after therapy assessed by gentle probing at 6 sites per tooth element

CONTACTS AND LOCATIONS:
Locations (1):
- CIR Dental School, Turin, Italy

IPD SHARING:
Plan to Share IPD: Undecided